CLINICAL TRIAL: NCT07195149
Title: Comparing High and lOw-dose asPirin With Dual anTIplatelet Therapy for Three Months Using prasUgrel and aSpirin Following Coronary Artery Bypass Grafting. (OPTIMUS-CABG Trial)
Acronym: OPTIMUS-CABG
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Dolnośląskie Centrum Chorób Serca im.prof. Zbigniewa Religi MEDINET Sp. z o.o. (Other)
Collaborators: Medical Research Agency, Poland (Other Government)
Responsible Party: Principal Investigator, Sleiman Sebastian Aboul-Hassan, Principal Investigator: Sleiman Sebastian Aboul-Hassan MD, PhD, Dolnośląskie Centrum Chorób Serca im.prof. Zbigniewa Religi MEDINET Sp. z o.o.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024/ABM/01/00016; 2025-521892-30-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-15; First posted 2025-09-26 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-11

CONDITIONS: Chronic Coronary Syndrome; Stable Coronary Artery Disease CAD
Keywords: DAPT; CABG; Prasugrel; Aspirin; CCS; Chronic coronary syndrome; Stable coronary artery disease
MeSH Terms: interventions — Aspirin; 2'-deoxythymidylyl-(3'-5')-2'-deoxyadenosine; Prasugrel Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Prasugrel 10 mg + Low Dose Aspirin 75 mg (Experimental)
  Interventions: Drug: DAPT (Low-Dose Aspirin 75 mg + Prasugrel 10 mg)
- Low-Dose Aspirin 75 mg (Active Comparator)
  Interventions: Drug: Low-Dose Aspirin 75 mg
- High-Dose Aspirin 300 mg (Active Comparator)
  Interventions: Drug: High-Dose Aspirin 300 mg

INTERVENTIONS:
Drug: High-Dose Aspirin 300 mg — High-dose Aspirin 300 mg once daily taken orally for three months
  Arms: High-Dose Aspirin 300 mg
Drug: DAPT (Low-Dose Aspirin 75 mg + Prasugrel 10 mg) — Drug: Prasugrel 10 mg
  Prasugrel 10 mg once daily taken orally for 3 months
  Drug: Low-Dose Aspirin
  75 mg once daily taken orally
  Arms: Prasugrel 10 mg + Low Dose Aspirin 75 mg
Drug: Low-Dose Aspirin 75 mg — Low-Dose Aspirin 75 mg once daily taken orally
  Arms: Low-Dose Aspirin 75 mg

SUMMARY:
The purpose of this study is to compare the effect of prasugrel plus low-dose aspirin versus high dose aspirin alone (300mg) and versus low dose aspirin alone (75 mg) in patients with chronic coronary disease undergoing coronary artery bypass grafting.

DETAILED DESCRIPTION:
This is a multicenter, randomized trial evaluating the effect of low-dose aspirin plus prasugrel versus low-dose ASA and versus high-dose ASA for three months, followed by low-dose ASA alone, on graft failure at 12 months in patients with stable coronary artery disease (chronic coronary syndrome) following a coronary artery bypass grafting.

ELIGIBILITY:
Inclusion Criteria:

A. Baseline (preoperative) inclusion criteria

1. Age >18 years
2. Primary isolated CABG patients with stable coronary artery disease (chronic coronary syndrome) planned for at least 2 grafts. Coronary artery disease will be defined as a stenosis ≥ 70% based on coronary angiography, a FFR value ≤ 0.80 or iFr value ≤0.89; a left main diameter stenosis ≥ 50%, left main IVUS MLA value ≤ 6 mm2, or equivalent OCT measurements will also be considered.
3. Ability to comply with all study procedures and follow-up procedures
4. Signed Informed Consent to participate in the study.

B. Operative inclusion criteria:

1. Intraoperative graft evaluation using transit time flow measurement in all grafts, normal flow in any graft is defined as mean graft flow > 15 mL/min with Pulsatility Index < 5
2. Left anterior descending artery grafted with internal thoracic artery
3. No intraoperative decision for hybrid revascularization due to incomplete revascularization (Percutaneous coronary intervention (PCI) of the ungrafted vessel)
4. No endarterectomy of the grafted vessel performed
5. Patient did not have any additional unplanned procedure (Ex. LAAC, Ablation, valve intervention, aortic intervention)

Exclusion Criteria:

A. Baseline (preoperative) exclusion criteria:

1. Cardiogenic shock
2. Patients with recent acute coronary syndrome (ACS) (<12 months)
3. Single vessel CABG
4. Patients with preoperative atrial fibrillation
5. Dialysis
6. Thrombocytopenia (platelet count < 100 000 platelets/uL)
7. Anemia (Hemoglobin level < 10 g/dL)
8. Severe liver failure Child-Pugh classification >4
9. Known, active infections with HIV, HBV, HCV, tuberculosis
10. Active malignant disease or history of malignancy within the past 5 years
11. Indication for DAPT (e.g. recent PCI or ACS or recent stents of peripheral arteries)
12. Indication for oral anticoagulant treatment 13 Indications for the use of methotrexate at a dose of 15 mg/week or more

14. Any contraindication for prasugrel or ASA 15. Planned additional cardiac or non-cardiac surgery within 12 months 16. Non-cardiac co-morbidity with life expectancy less than 12 months 17. History of any bleeding complications due to the use of DAPT 18. History of intracranial bleeding 19. History of gastro-intestinal bleeding 20. Pregnancy or breastfeeding 21. Lack of compliance with the use of a highly effective method of birth control 22. Planned coronary endarterectomy 23. Severe impaired renal function (eGFR <40mL/min/1.73 m2).

B. Postoperative and prior randomization exclusion criteria:

1. Perioperative cardiogenic shock
2. Intraoperative death or death prior randomization
3. Myocardial infarction within 12-24 hours following CABG or prior randomization
4. Ischemic or hemorrhagic stroke within 12-24 hours following CABG or prior randomization
5. Any postoperative complication that may increase patients' risk with DAPT
6. Atrial Fibrillation prior randomization
7. Gastro-intestinal bleeding prior randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1703 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2030-04-30 (Estimated); Study Completion 2030-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of graft failure: DAPT vs Low-Dose Aspirin and DAPT vs High-Dose Aspirin | 12 months
  Incidence of graft failure defined according to Fitzgibbon classification (Fitzgibbon Class B + O) 12 months after the randomization following CABG in patients with DAPT (prasugrel 10mg/day + low dose aspirin 75mg/day) versus high-dose aspirin (300mg/day) and in patients with DAPT (prasugrel 10mg/day + low dose aspirin 75mg/day) vs low-dose aspirin (75mg/day)

SECONDARY OUTCOMES:
Key secondary outcome: Incidence of graft failure: High-Dose Aspirin vs Low-Dose Aspirin | 12 months
  Incidence of graft failure defined according to Fitzgibbon classification (Fitzgibbon Class B + O) 12 months after the randomization following CABG in patients with high-dose aspirin (300mg/day) vs low-dose aspirin (75mg/day)
investigatigating the effect of DAPT versus low-dose aspirin, DAPT versus high-dose aspirin and low-dose aspirin versus high-dose aspirin on the 12-month risk of ischemic events after CABG | 12 months
  Major adverse cardiac and cerebral events (MACCE) is a composite endpoint to be compared between groups defined as composite of:
  1. All-cause mortality
  2. Incidence of myocardial infarction
  3. Incidence of stroke
  4. Incidence of repeat revascularization
Investigatigating the effect of DAPT versus low-dose aspirin, DAPT versus high-dose aspirin and low-dose aspirin versus high-dose aspirin on the 12-month risk of bleeding events after CABG | 12 months
  Incidence of bleeding within 12 months after randomization following CABG procedure according to the Bleeding Academic Research Consortium (BARC) type 2, 3 or 5
Investigatigating the effect of DAPT versus low-dose aspirin, DAPT versus high-dose aspirin and low-dose aspirin versus high-dose aspirin on quality of life at 6 and 12 months after CABG. | 12 months
  Quality of life will be assessed using quality of life questionnaires at baseline, 6 and 12 months after randomization following CABG procedure and will be evaluated using The Seattle Angina Questionnaire - 7 (SAQ-7) and Short-form-12 health survey questionnaire (SF-12)
investigatigating the effect of DAPT versus low-dose aspirin, DAPT versus high-dose aspirin and low-dose aspirin versus high-dose aspirin on the 60-month risk of ischemic events after CABG | 60 months
  Major adverse cardiac and cerebral events (MACCE) is a composite endpoint to be compared between groups defined as composite of:
  1. All-cause mortality
  2. Incidence of myocardial infarction
  3. Incidence of stroke
  4. Incidence of repeat revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Sleiman Sebastian Aboul-Hassan, MD, PhD, Principal Investigator — Zbigniew Religa Heart Center "Medinet"
Locations (18):
- Poland (18):
  - University Clinical Hospital in Bialystok, Bialystok
  - Nicolaus Copernicus University Ludwik Rydygier Collegium Medicum in Bydgoszcz, Bydgoszcz
  - Medical University of Gdansk, Gdansk
  - Regional Specialist Hospital in Grudziadz, Grudziądz
  - Upper-Silesian Heart Center, Katowice
  - John Paul II Hospital, Krakow
  - Medical University of Lodz, Lodz
  - Zbigniew Religa Heart Center "Medinet", Nowa Sól
  - Provincial Specialist Hospital in Olsztyn, Olsztyn
  - Institute of Medical Sciences in Opole, Opole
  - J. Struś Hospital, Poznan
  - Poznan University of Medical Sciences, Poznan
  - Pomeranian Medical University, Szczecin
  - Central Clinical Hospital of the Ministry of Interior and Administration, Warsaw
  - Medicover Hospital, Warsaw
  - Wroclaw Medical University, Wroclaw
  - Zbigniew Religa Heart Center "Medinet", Wroclaw
  - Silesian Centre for Heart Diseases in Zabrze, Zabrze

IPD SHARING:
Plan to Share IPD: No